CLINICAL TRIAL: NCT05622604
Title: The Effect of Religious Practices on Mental and Spiritual Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biola University (Other)
Responsible Party: Principal Investigator, Todd Hall, Professor, Biola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F22-011
Record Dates: First submitted 2022-11-08; First posted 2022-11-18 (Actual); Results first posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Stress

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three conditions. Condition 1 is the control condition (i.e., no intervention condition). In Condition 2, participants will be given a free subscription to the Pray.com app and will be directed to use the app five days per week (i.e., autonomous use condition). In Condition 3, participants will be given a free subscription to the Pray.com app and will be directed to listen to a meditation prayer five days per week (i.e., meditative prayer condition).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no intervention condition (No Intervention): no intervention
- autonomous use condition (Experimental): Participants will be given a free subscription to the Pray.com app and will be directed to use the app five days per week.
  Interventions: Behavioral: pray.com app (autonomous use)
- meditative prayer condition (Experimental): Participants will be given a free subscription to the Pray.com app and will be directed to listen to a meditation prayer five days per week.
  Interventions: Behavioral: pray.com app (meditative prayer condition)

INTERVENTIONS:
Behavioral: pray.com app (autonomous use) — Participants will be given a free subscription to the Pray.com app and will be directed to use the app five days per week.
  Arms: autonomous use condition
Behavioral: pray.com app (meditative prayer condition) — Participants will be given a free subscription to the Pray.com app and will be directed to listen to a meditation prayer five days per week.
  Arms: meditative prayer condition

SUMMARY:
The goal of this clinical trial is to test the effects of using a religious mobile app (i.e., Pray.com) in participants who have high levels of stress. The main question it aims to answer is:

•What are the effects of using Pray.com on stress in individuals who report high levels of stress?

Participants will complete measures at baseline (i.e., Time 1), four-weeks (i.e., Time 2), and eight weeks (i.e., Time 3). Participants will be randomly assigned one of three conditions: (1) autonomous use (directed to use the app daily), (2) meditative prayer condition (directed to use this feature of the app daily), or (3) wait-list control condition.

DETAILED DESCRIPTION:
Participants (N = 300) will be adults recruited through social media and faith-based organizations. Participants will first complete a brief screener to determine eligibility for the study.

Eligible participants will be invited to participate in the study. Participants will read an informed consent document that will give information about the study and their rights as participants. Participants will be given the opportunity to contact the research team and ask questions. If they agree to participate, participants will be randomly assigned to one of three conditions. Condition 1 is the control condition (i.e., no intervention condition). In Condition 2, participants will be given a free subscription to the Pray.com app and will be directed to use the app five days per week (i.e., autonomous use condition). In Condition 3, participants will be given a free subscription to the Pray.com app and will be directed to listen to a meditation prayer five days per week (i.e., meditative prayer condition). Participants will receive periodic reminders on their phone if they have not used the app.

All participants will fill out a series of online questionnaires monthly for a two-month time-period (i.e., Baseline / Time 1, Time 2, and Time 3). Participants will receive a link from the research team when it is time for them to fill out their questionnaire via a secure online data collection portal. After finishing the study, participants will be debriefed and given the opportunity to ask questions about their participation.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* own a smart phone and be willing to download a mobile app
* willing to engage in a Christian practice on a mobile app
* score of 14 or greater on the Perceived Stress Scale (indicating at least a moderate level of stress)

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Hall, PhD, Principal Investigator — Biola University
Locations (1):
- Biola University, La Mirada, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial protocol enrollment was 312. However, 120 participants were removed from the study due to suspicions of poor data quality and invalid responses (e.g., same internet protocol addresses across multiple participants, unusual responses), leaving 192 valid participants.
Period: Overall Study
Arm/Group | no Intervention Condition | Autonomous Use Condition | Meditative Prayer Condition
Started | 80 | 56 | 56
Completed | 58 | 33 | 44
Not Completed | 22 | 23 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | no Intervention Condition | Autonomous Use Condition | Meditative Prayer Condition | Total
Number analyzed (Participants) | 80 | 56 | 56 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 79 | 55 | 56 | 190
  >=65 years | 1 | 1 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.46 (11.17) | 36.54 (12.13) | 36.45 (10.48) | 36.48 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 39 | 37 | 129
  Male | 27 | 17 | 19 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasion | 65 | 41 | 44 | 150
  Black or African American | 3 | 12 | 6 | 21
  Asian or Asian American | 8 | 1 | 2 | 11
  Latina/Latino American | 2 | 1 | 2 | 5
  Biracial or multiracial | 1 | 1 | 1 | 3
  Other | 1 | 0 | 1 | 2
Perceived Stress Scale -10 [Mean (Standard Deviation); unit: units on a scale] | 3.39 (.62) | 3.12 (.52) | 3.19 (.63) | 3.30 (.60)
Hospital Anxiety and Depression Scale [Mean (Standard Deviation); unit: units on a scale]
  Anxiety | 1.65 (.45) | 1.52 (.47) | 1.57 (.49) | 1.59 (.47)
  Depression | 1.03 (.53) | .99 (.56) | .95 (.52) | 1.00 (.54)
Mindful Attention and Awareness Scale [Mean (Standard Deviation); unit: units on a scale] | 3.69 (.77) | 3.63 (.80) | 3.62 (.71) | 3.66 (.76)
Copenhagen Burnout Inventory [Mean (Standard Deviation); unit: units on a scale] | 3.58 (.67) | 3.50 (.69) | 3.48 (.67) | 3.53 (.68)
Pittsburgh Sleep Quality Index [Mean (Standard Deviation); unit: units on a scale] | 17.96 (3.47) | 17.44 (3.17) | 17.86 (3.04) | 17.82 (3.26)
Religious Community Inventory [Mean (Standard Deviation); unit: units on a scale] | 3.85 (.79) | 3.77 (.85) | 3.78 (.84) | 3.81 (.82)
Spiritual Well-Being Scale [Mean (Standard Deviation); unit: units on a scale] | 4.51 (.84) | 4.56 (.68) | 4.54 (.76) | 4.53 (.78)
Satisfaction with Life Scale [Mean (Standard Deviation); unit: units on a scale] | 4.06 (1.39) | 4.18 (1.15) | 4.32 (1.43) | 4.15 (1.35)
Productivity [Mean (Standard Deviation); unit: units on a scale] | 3.33 (1.05) | 3.53 (.81) | 3.54 (.84) | 3.45 (.93)

OUTCOME MEASURES:

1. Primary Outcome: Perceived Stress Scale
Description: minimum value: 0, maximum value: 4, higher average item scores indicate higher levels of stress (i.e., worse outcome)
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | no Intervention Condition | Autonomous Use Condition | Meditative Prayer Condition
Number analyzed (Participants) | 58 | 33 | 44
units on a scale | 2.79 (.65) | 2.71 (.57) | 2.65 (.65)

2. Secondary Outcome: Hospital Anxiety and Depression Scale
Description: minimum value: 0, maximum value: 3, higher average item scores indicate higher levels of anxiety/depression (i.e., worse outcome)
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | no Intervention Condition | Autonomous Use Condition | Meditative Prayer Condition
Number analyzed (Participants) | 58 | 33 | 44
units on a scale
  Anxiety | 1.17 (.49) | 1.00 (.46) | .95 (.46)
  Depression | .66 (.50) | .63 (.56) | .59 (.46)

3. Secondary Outcome: Mindful Attention Awareness Scale
Description: minimum value: 1, maximum value: 6, higher average item scores indicate higher levels of mindfulness (i.e., better outcome)
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | no Intervention Condition | Autonomous Use Condition | Meditative Prayer Condition
Number analyzed (Participants) | 58 | 33 | 44
units on a scale | 3.14 (.96) | 2.87 (.75) | 2.89 (.96)

4. Secondary Outcome: Copenhagen Burnout Inventory--personal Subscale
Description: minimum value: 0, maximum value: 4, higher average item scores indicate higher levels of burnout (i.e., worse outcome)
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | no Intervention Condition | Autonomous Use Condition | Meditative Prayer Condition
Number analyzed (Participants) | 58 | 33 | 44
units on a scale | 2.93 (.91) | 2.80 (.72) | 2.76 (.79)

5. Secondary Outcome: Pittsburgh Sleep Quality Inventory
Description: Each component score of the scale ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a total score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | no Intervention Condition | Autonomous Use Condition | Meditative Prayer Condition
Number analyzed (Participants) | 58 | 33 | 44
score on a scale | 13.43 (3.13) | 13.21 (2.88) | 13.55 (2.91)

6. Secondary Outcome: Religious Commitment Inventory
Description: minimum value: 1, maximum value: 5, higher average item scores indicate higher levels of religious commitment (i.e., better outcome)
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | no Intervention Condition | Autonomous Use Condition | Meditative Prayer Condition
Number analyzed (Participants) | 58 | 33 | 44
units on a scale | 4.06 (.74) | 3.85 (.93) | 4.07 (.76)

7. Secondary Outcome: Spiritual Well-Being Scale
Description: minimum value: 1, maximum value: 6, higher average item scores indicate higher levels of spiritual well-being (i.e., better outcome)
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | no Intervention Condition | Autonomous Use Condition | Meditative Prayer Condition
Number analyzed (Participants) | 58 | 33 | 44
units on a scale | 4.89 (.79) | 4.79 (1.02) | 4.85 (.77)

8. Secondary Outcome: Satisfaction With Life Scale
Description: minimum value: 1, maximum value: 7, higher average item scores indicate higher levels of satisfaction with life (i.e., better outcome)
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | no Intervention Condition | Autonomous Use Condition | Meditative Prayer Condition
Number analyzed (Participants) | 58 | 33 | 44
units on a scale | 4.92 (1.35) | 4.86 (1.32) | 4.91 (1.31)

9. Secondary Outcome: Productivity
Description: Participants' level of productivity was measured by three items (Vogel et al., 2022): Participants were asked to rate their responses on a scale from 1 = strongly disagree to 5 = strongly agree. Participants' mean responses were calculated, with higher scores indicating higher perceived efficiency and productivity
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | no Intervention Condition | Autonomous Use Condition | Meditative Prayer Condition
Number analyzed (Participants) | 58 | 33 | 44
units on a scale | 3.86 (.82) | 3.86 (.89) | 4.00 (.86)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | no Intervention Condition | Autonomous Use Condition | Meditative Prayer Condition
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/80 | 0/56 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT05622604/Prot_SAP_ICF_000.pdf